CLINICAL TRIAL: NCT00177515
Title: Preventive Health Education for Women of Reproductive Age
Brief Title: Computer-assisted Preventive Health Education for Women of Reproductive Age in Urgent Care Settings
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Eleanor Schwarz, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: H2582-25916-01A
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Preconception Care
Keywords: emergency contraception; folic acid; education; preventive health

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Computerized counseling about Emergency Contraception
  Interventions: Behavioral: "video doctor," computer module
- 2 (Active Comparator): Computerized counseling about peri-conception folate
  Interventions: Behavioral: "video doctor," computer module

INTERVENTIONS:
Behavioral: "video doctor," computer module — computerized counseling about emergency contraception and peri-conception folate
  Other Names: EC and folate arms

SUMMARY:
The purpose of this study is to determine whether "video doctor" programs can effectively deliver preventive health messages to women of reproductive age while they wait to be seen in urgent care settings. In this study, the specific hypotheses being tested are: 1) is the video doctor program effective in improving women's knowledge about emergency contraception, and 2) is the video doctor program effective in improving women's knowledge about the importance of folate.

DETAILED DESCRIPTION:
We will randomly assign participants to interact with one of two "video doctor" programs which have been been developed to convey messages appropriate for women of reproductive age.

The "video doctor" is an actress (not UCSF staff) following a script that has been designed through interdisciplinary collaboration here at UCSF. These particular video programs have not been used before, but similar ones have been studied and shown to be effective by Dr. Gerber in providing patients with information about how to decrease sexual risks and the harms of alcohol and drug use. Before interacting with the "video doctor" program, we will assess participants baseline knowledge of the importance of peri-conception folate and the option of emergency contraception. Participants will then interact with their "video doctor" and be provided with a free sample of the pills their video doctor discussed.

The first "video doctor" will educate women about the ability of folate to reduce birth defects. The discovery that peri-conception folate supplementation significantly decreases rates of neural tube defects has inspired multiple educational campaigns. However, recent work has shown that knowledge of the benefits of folate remains low, especially among minority populations.

The second "video doctor" message will inform women of the option of emergency contraception. Emergency contraception using high doses of progesterone has been shown to reduce the risk of pregnancy to less than 2% when used up to five days after a condom failure or an episode of unprotected sex.

This medication is not teratogenic and will not cause a miscarriage if used by a woman who does not know she is pregnant. Use of emergency contraception poses no long-term health risks to women and is available over-the-counter in seven European countries. Prior studies in family planning clinics , as well as the post-partum setting have shown that education about and advance provision of emergency contraceptive pills can increase knowledge and appropriate use of these pills, without adversely affecting sexual risk taking or other health behaviors. However, knowledge of emergency contraception remains limited, leading some to call it America's "best kept secret." Participants will be contacted by phone six months after interacting with the "video doctor" and asked to provide information about their use of folate and/or emergency contraception. One year after interacting with the "video doctor" participants will be contacted again and asked to provide further information about their use of folate and/or emergency contraception.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 year old English-speaking women

Exclusion Criteria:

* current pregnancy
* history of tubal ligation
* hysterectomy
* partner with a vasectomy
* no sex with men
* will not be able to be reached by telephone in 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 446 (Actual)
Dates: Start 2005-03; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Use of Emergency Contraception | 7 months
Use of Folate supplements | 7 months

SECONDARY OUTCOMES:
Access to Emergency Contraception at home | 7 months
Knowledge of emergency contraception | 7 months
Knowledge of the benefits of folate supplementation | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor B Schwarz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Schwarz EB, Gerbert B, Gonzales R. Computer-assisted provision of emergency contraception a randomized controlled trial. J Gen Intern Med. 2008 Jun;23(6):794-9. doi: 10.1007/s11606-008-0609-x. Epub 2008 Apr 9. PMID 18398664
- [Derived] Schwarz EB, Sobota M, Gonzales R, Gerbert B. Computerized counseling for folate knowledge and use: a randomized controlled trial. Am J Prev Med. 2008 Dec;35(6):568-71. doi: 10.1016/j.amepre.2008.06.034. PMID 19000845
- See also: Computerized Counseling for Folate Knowledge and Use — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2593421/